CLINICAL TRIAL: NCT03578848
Title: A Randomized Controlled Trial Comparing Unattended Automated Office Blood Pressure vs. Home Blood Pressure vs. Central Blood Pressure Monitoring for the Management of Hypertension
Brief Title: Guiding Hypertension Management Using Different Blood Pressure Monitoring Strategies
Acronym: GYMNs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018-05-009A
Record Dates: First submitted 2018-06-04; First posted 2018-07-06 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
Keywords: blood pressure monitoring; sphygmomanometer
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: BP will be taken simultaneously from both upper arms by an oscillometric BP monitor. Subjects with SBP Differences between both arms more than 5 mmHg will be excluded. For the unattended automated BP (uAOBP) and central BP (CBP), the measurements will be conducted in a quiet room without the presence of clinical personnel. Simultaneously, the central BP will be measured in the other upper arm. The determination of the right or left upper arm for uAOBP or central BP will be made in a random order by computer generated random codes before the enrollment. As for the home BP measurements, a validated device will be provided for all subjects allocated to the home BP arm to measure their BP at home. Subjects are requested to take BP in the morning and afternoon before meals for 7 consecutive days before the scheduled clinical visits. BP in the first day of the measurements will be discarded and an average of home BP will be generated and provided for clinicians to guide their treatment.
Who Masked: Participant, Care Provider
Masking Description: Each patient will be randomly assigned, using a standard computer protocol at the General Clinical Research Center, Taipei Veterans General Hospital, Taipei, Taiwan, to intervention in a 1:1:1 ratio to home BP, uAOBP, or central BP using sealed opaque envelopes (sequentially numbered). The study coordinator will oversee the enrollment and intervention assignment and keep allocation concealment. The caring physicians will remain blinded to the allocation by providing them with the measured BP values through a standardized report form without the knowledge of the used BP monitoring devices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- uAOBP & Home BP (Active Comparator): On the scheduled visits, the uAOBP and Home BP will be measured before meeting doctors and provided for clinicians to adjust patients' medication according to practice guideline.
  Interventions: Device: uAOBP; Device: Home BP
- CBP & Home BP (Experimental): On the scheduled visits, the CBP and Home BP will be measured before meeting doctors and provided for clinicians to adjust patients' medication according to practice guideline.
  Interventions: Device: Home BP; Device: CBP

INTERVENTIONS:
Device: uAOBP — For the uAOBP and CBP, the measurements will be conducted in a quiet room without the presence of clinical personnel. Patients will be seated in a quiet room without talking and taken as an average of 3 measurements with an automated device (HEM-907, Omron Healthcare, Lake Forest, IL) that has been preset to wait 5 minutes before measurements. Simultaneously, the central BP will be measured in the other upper arm. (WatchBP Office Central; Microlife AG, Widnau, Switzerland). The determination of the right or left upper arm for uAOBP or central BP will be made in a random order by computer generated random codes before the enrollment.
  Arms: uAOBP & Home BP
Device: Home BP — As for the home BP measurements, a validated device (WatchBP Home; Microlife AG, Widnau, Switzerland) will be provided for all subjects allocated to the home BP arm to measure their BP at home. Subjects are requested to take BP in the morning (within 2 hours after awakening) and afternoon before meals for 7 consecutive days before the scheduled clinical visits. BP in the first day of the measurements will be discarded and an average of home BP (all BP reading and BP in the morning and in the afternoon) will be generated and provided for clinicians to guide their treatment.
Device: CBP — For the uAOBP and CBP, the measurements will be conducted in a quiet room without the presence of clinical personnel. Patients will be seated in a quiet room without talking and taken as an average of 3 measurements with an automated device (HEM-907, Omron Healthcare, Lake Forest, IL) that has been preset to wait 5 minutes before measurements. Simultaneously, the central BP will be measured in the other upper arm. (WatchBP Office Central; Microlife AG, Widnau, Switzerland). The determination of the right or left upper arm for uAOBP or central BP will be made in a random order by computer generated random codes before the enrollment.
  Arms: CBP & Home BP

SUMMARY:
Patients with uncontrolled or newly diagnosed hypertension will be randomized to have hypertension management decisions made on the basis of the unattended automated blood pressure (uAOBP) , home BP, and central BP monitoring. This study evaluates the optimal guiding strategy for hypertension will help define which BP monitoring is the most effective strategy to guide the clinical management of hypertension.

DETAILED DESCRIPTION:
The traditional BP used for clinical practice, the office BP, is usually measured in a busy and hurry clinical environment, and interfered by the well-known confounding whitecoat effect. As such, unattended automated office BP monitoring (uAOBP) has been proposed as an effective solution and further promoted by Canadian physicians.

Nonetheless, out-of-office BP, home BP and ambulatory BP, remains the methodology of recommendation for the detection of whitecoat effect, and its prognostic value has been demonstrated to be superior to the traditional office BP. Home BP monitoring, with its ability to detect morning and masked hypertension and a better tolerability than ambulatory BP monitoring for long-term use, can therefore be considered as a strategy of choice to replace office BP monitoring for guiding hypertension management.

Moreover, BP measurements in the peripheral arteries cannot serve as direct substitutes for their central counterparts because of the long-recognized differences of blood pressure (BP) waveforms and values between the central aorta and peripheral arterial system. Thus, if the decisions on medication adjustment are made solely based brachial BP, there could be a considerable risk of over- or undertreatment.

Considering that there are many better strategies for guiding hypertension management than traditional office BP, there is an apparent need for investigating their comparative effectiveness and safety in the management of hypertension. The investigators hypothesized that home BP may be non-inferior to AOBP and central BP-guided intervention in reducing ambulatory BP and designed the present randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 90 years of age
* nonpregnant
* receiving antihypertensive therapy for uncomplicated essential hypertension and taking ≥1 but ≤ 2 types antihypertensive drugs (to rule out complicated or resistant hypertension) or hypertension newly diagnosed by uAOBP (uAOBP >130 mmHg at screening visit)

Exclusion Criteria:

* Poor adherence to medication
* unable to conduct self-measurement blood pressure
* history of polycystic kidney disease
* congestive heart failure (a recent assessment of left ventricular ejection fraction < 40% prior to screening visit)
* chronic kidney disease with estimated glomerular filtration rate < 30 mL/min/1.73m2 (MDRD) at screening visit
* a recent document of severely abnormal left ventricular mass index (>59 g/m2.7 in women and >64 g/m2.7 in men) prior to screening visit
* secondary causes of hypertension
* uncontrolled hypertension (uAOBP >180/100 mm Hg at screening visit)
* history of severe aortic valve disease
* history of upper limb obstructive atherosclerosis
* history of atrial fibrillation
* BP Differences more than 5 mmHg between both arms at screening visit

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
24 hour mean ambulatory systolic blood pressure | 3 months
  The change of 24 hour mean ambulatory systolic blood pressure (SBP)

SECONDARY OUTCOMES:
24 hour mean ambulatory diastolic blood pressure | 3 months
  The change of 24 hour mean ambulatory diastolic blood pressure (DBP)
left ventricular mass | 12 months
  decrease of left ventricular mass
SBP and DBP | 12 months
  change of SBP/DBP measured by uAOBP monitoring, home BP monitoring, or central BP monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Min Cheng, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Cheng HM, Sung SH, Chen CH, Yu WC, Yang SM, Guo CY, Chuang SY, Chiang CE. Guiding Hypertension Management Using Different Blood Pressure Monitoring Strategies (GYMNs study): comparison of three different blood pressure measurement methods: study protocol for a randomized controlled trial. Trials. 2019 May 10;20(1):265. doi: 10.1186/s13063-019-3366-8. PMID 31077229

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT03578848/Prot_SAP_ICF_000.pdf